CLINICAL TRIAL: NCT07061002
Title: Evaluation of Recruitment Effectiveness in Patients With Obstructive Sleep Apnea Syndrome Using Lung Ultrasound
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Münevver Kayhan, Lecturer, Istanbul University - Cerrahpasa
Allocation: Not Applicable | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: ctf-osas-recruitment-01
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Atelectasis; Lung Ultrasonography Score; Recruitment
Keywords: Postoperative Pulmonary Atelectases; lung ultrasound score; recruitment maneuver
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: After participants are enrolled and informed consent is obtained, they will be randomly assigned to one of three groups in a 1:1:1 ratio using a computer-generated randomization list prepared by an independent anesthesiologist who is not involved in the intervention. Allocation concealment will be ensured using sequentially numbered, opaque, sealed envelopes for each patient. To maintain double blinding, both the patients and the researchers responsible for postoperative evaluations (including those performing lung ultrasound and clinical follow-ups) will remain unaware of group assignments. The intraoperative team responsible for performing the intervention will only carry out the assigned procedure and will not be involved in data collection, evaluation, or analysis. Group assignments will be documented separately and kept confidential until the study is completed and data analysis is finalized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1- control (No Intervention): The patient will be ventilated throughout the surgery by applying 5 cmH2O post expiratory positive end-expiratory pressure. Lung ultrasound will be performed on the patients before surgery, 5 minutes after mechanical ventilation after orotracheal intubation, at the end of surgery and 5 minutes after extubation. The lung will be evaluated in 8 regions. These will be evaluated as upper and lower in the mid-clavicular line, upper and lower in the anterior axillary line, upper and lower in the posterior axillary line and Plaps point. It will be evaluated by calculating the modified Lung Ultrasound Score (LUSS) to detect ventilation loss. Higher scores in LUSS indicate more severe ventilation loss. The degree of deaeration will be evaluated between 0 and 3. , 0 less than 3 B line; ≥3 B lines indicate 1, greater than 5 and confluent B lines indicate 2, and multiple confluent B lines or multiple subpleural consolidations separated by a thickened or irregular pleural line indicate 3.
- Group 2 (Active Comparator): The ventilation strategy of the patients in this group will be the same as in group 1. In contrast, just before extubation, the patients in this group will be given 6 breaths with a tidal volume of 2 times the vital capacity, an inspiratory/expiratory ratio of 1/1 and a lung plateau pressure of < 35 cmH2O, and a recruitment maneuver will be performed at the end of the surgery. All patients will undergo lung ultrasound in the defined lung zones and at the specified times, as described in group 1, and a modified Lung Ultrasound score will be evaluated.
  Interventions: Other: Lung Recruitment Maneuver
- Group 3 (Active Comparator): The ventilation strategy of the patients in this group will be the same as in group 1. In addition to positive end-expiratory pressure, the patient will be placed in the right and then left lateral decubitus position before extubation at the end of the surgery and a recruitment maneuver will be performed by giving 6 breaths in each position with a tidal volume twice the vital capacity, a 1/1 inspiratory/expiratory ratio and a lung plateau pressure < 35 cmH2O. All patients will undergo lung ultrasound in defined lung regions and at specified times, as defined in group 1, and a modified Lung Ultrasound score will be evaluated.
  Interventions: Other: Positional Lung Recruitment Maneuver

INTERVENTIONS:
Other: Lung Recruitment Maneuver — Lung Recruitment Maneuver (LRM) is a method that allows the alveoli to reopen by applying high positive pressure in order to prevent or treat alveolar collapse (atelectasis) that develops during or after anesthesia. LRM improves oxygenation by increasing functional residual capacity. Clinical studies have shown that LRM increases oxygenation levels, reduces areas of atelectasis, and shortens hospital stay. In this study, the effects of different recruitment maneuvers on postoperative atelectasis will be evaluated. In this group, just before extubation, the patients in this group will be given 6 breaths with a tidal volume of 2 times the vital capacity, an inspiratory/expiratory ratio of 1/1 and a lung plateau pressure of < 35 cmH2O, and a recruitment maneuver will be performed at the end of the surgery.
  Arms: Group 2
Other: Positional Lung Recruitment Maneuver — Lung Recruitment Maneuver (LRM) is a method that allows the alveoli to reopen by applying high positive pressure in order to prevent or treat alveolar collapse (atelectasis) that develops during or after anesthesia. LRM improves oxygenation by increasing functional residual capacity. Clinical studies have shown that LRM increases oxygenation levels, reduces areas of atelectasis, and shortens the length of hospital stay. In this study, the effects of different recruitment maneuvers on postoperative atelectasis will be evaluated. Patients in this group will be placed in the right and then left lateral decubitus position before extubation at the end of surgery and a recruitment maneuver will be performed by giving 6 breaths in each position, with a tidal volume twice the vital capacity, a 1/1 inspiratory/expiratory ratio, and a lung plateau pressure < 35 cmH2O.
  Arms: Group 3

SUMMARY:
Patients with obstructive sleep apnea syndrome are at higher risk for respiratory complications after surgery. Oxygen depletion and respiratory distress are common in patients with obstructive sleep apnea syndrome. In this study, the effectiveness of the recruitment maneuver applied in the postoperative period will be investigated via lung ultrasound. Recruitment is a technique performed to improve the oxygen levels of patients. Patients diagnosed with obstructive sleep apnea syndrome between the ages of 18-65 will be included in the study and anesthesia and surgical procedures will be followed. The aim of the study is to compare the pulmonary complication rates between patients who underwent recruitment and those who did not, and to examine the effects of factors such as age and gender on these complications via lung ultrasound.

DETAILED DESCRIPTION:
The effect of the recruitment maneuver applied in the postoperative period on lung ventilation and atelectasis will be investigated via lung ultrasound. Recruitment is a technique performed to improve the oxygen levels of patients. Patients diagnosed with obstructive sleep apnea between the ages of 18-65 will be included in the study. The aim of the study is to compare atelectasis rates, pleural fascial fluid accumulation, lung compliance, pneumothorax findings between patients who underwent and did not undergo recruitment with lung ultrasound. In addition, to examine the effects of factors such as age and gender on these complications with lung ultrasound. Our study is a prospective, single-center, control group clinical trial to be conducted on patients diagnosed with obstructive sleep apnea syndrome (OSA). Patients between the ages of 18-65, classified as American Society of Anesthesia I-III, and diagnosed with Obstructive Sleep Apnea (polysomnography or STOP-BANG score ≥3) will be included in the study. Written informed consent will be obtained from the patients before the surgical procedure. Patients to be excluded from the study will include American Society of Anesthesia class IV and above patients, those with a history of neuromuscular disease, patients requiring cardiac surgery, and patients requiring urgent surgical intervention.

Patients will be randomly divided into three groups by computer-based program: Group 1: A fixed 5 cmH2O post expiratory positive end-expiratory pressure will be applied. Group 2: In addition to the fixed positive end-expiratory pressure, a recruitment maneuver will be performed at the end of surgery before extubation by giving 6 breaths with a tidal volume at 2 times the vital capacity, an inspiration/expiration ratio of 1/1, and a lung plateau pressure of < 35 cmH2O. Group 3: In addition to the fixed positive end-expiratory pressure, a recruitment maneuver will be performed at the end of surgery by giving 6 breaths in the right and left lateral decubitus positions before extubation. All patients' preoperative demographic data, apnea device usage, chest X-ray, total anesthesia duration, surgical duration, drugs used and their doses, ventilation parameters (tidal volume, positive end-expiratory pressure, airway peak pressure), fluid balance, surgical procedure type, patient position data will be recorded. Hemodynamic parameters, oxygen, respiratory exercise and bronchodilator requirements of patients taken to the recovery unit will be recorded. Lung A line and B line scores will be evaluated separately as 8 zones while performing lung ultrasonography of all patients. Plasm points, air bronchogram findings, pleural sliding movements will be recorded for each zone. In these follow-ups, saturation, hemodynamic parameters, respiratory exercise, bronchodilator requirement, intubation requirement, unplanned intensive care admission, hospital stay duration will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65
* American Society of Anesthesia I-III
* Patients with consent to participate
* Patients with preoperative OSA diagnosis (polysomnography or STOP-BANG≥3)

Exclusion Criteria:

* American Society of Anesthesia >IV
* Patients planned for postoperative intensive care follow-up 3. Cardiac surgery
* Anesthesia outside the operating room
* History of neuromuscular disease
* Emergency surgical application
* Invasive airway surgeries (pharynx, larynx)
* Lung surgeries (pneumonectomy, lobectomy, etc.) 9. Presence of pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-07-25 (Estimated); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
pulmonary complications underwent recruitment maneuver | 10 minutes before the start of surgery until 10 minutes after the end of surgery
  The primary outcome of the study was to compare the pulmonary complication rates between patients who underwent the recruitment maneuver and those who did not by lung ultrasound. Pulmonary complications were assessed by using the modified lung ultrasound score (LUSS). Higher scores on the LUSS indicated more severe ventilation loss. The degree of deaeration was assessed from 0 to 3. , Less than 3 B lines; ≥3 B lines were rated as 1, greater than 5 and confluent B lines were rated as 2, and multiple confluent B lines separated by a thickened or irregular pleural line or multiple subpleural consolidations were rated as 3.

SECONDARY OUTCOMES:
Pulmonary Complications with Different Recruitment Maneuver Techniques | 10 minutes before the start of surgery until 10 minutes after the end of surgery
  The secondary outcome is to compare the pulmonary complication rates between patients who received different recruitment maneuver techniques. To compare the postoperative pulmonary complication rates of parameters such as age, gender, and body mass index. Pulmonary complications will be assessed by performing the modified lung ultrasound score (LUSS). Higher scores on the LUSS indicate more severe ventilation loss. The degree of deaeration will be assessed from 0 to 3. , Less than 3 B lines; ≥3 B lines indicate 1, greater than 5 and confluent B lines indicate 2, and multiple confluent B lines separated by thickened or irregular pleural lines or multiple subpleural consolidations indicate 3.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Cigdem Tutuncu, Professor, Study Chair — Istanbul University-Cerrahpasa, Cerrahpasa Medicine of Faculty; Munevver Kayhan, Lecturer Doctor, Principal Investigator — Istanbul University-Cerrahpasa, Cerrahpasa Medicine of Faculty; Pinar Kendigelen, Professor Doctor, Principal Investigator — Istanbul University-Cerrahpasa, Cerrahpasa Medicine of Faculty
Locations (1):
- Istanbul University-Cerrahpasa, Cerrahpasa Medicine of Faculty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Touw HR, Schuitemaker AE, Daams F, van der Peet DL, Bronkhorst EM, Schober P, Boer C, Tuinman PR. Routine lung ultrasound to detect postoperative pulmonary complications following major abdominal surgery: a prospective observational feasibility study. Ultrasound J. 2019 Sep 16;11(1):20. doi: 10.1186/s13089-019-0135-6. PMID 31523784
- [Result] Canet J, Hardman J, Sabate S, Langeron O, Abreu MG, Gallart L, Belda J, Markstaller K, Pelosi P, Mazo V. PERISCOPE study: predicting post-operative pulmonary complications in Europe. Eur J Anaesthesiol. 2011 Jun;28(6):459-61. doi: 10.1097/EJA.0b013e328344be2d. No abstract available. PMID 21544025